CLINICAL TRIAL: NCT07048756
Title: Enhancing the Efficacy of Psychotherapeutic Imagery Techniques: A Randomized Controlled Trial
Brief Title: Psychotherapeutic Imagery Techniques
Acronym: JM2019a
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Jaroslaw Michalowski, Professor, University SWPS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SONATA_BIS_JM2019a
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Fear of Failure
Keywords: Imagery Rescripting; Imagery Exposure; Schema Therapy; Compassion Focused Therapy; Fear of Failure; Disruption of Reconsolidation; Skin Conductance Level

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Imagery Rescripting (ImRs) (Experimental): Before treatment each participant took part in 2 imagery sessions during which a cognitive-behavioral therapist (CBT) asked him/her to recall 3 events of being criticized for failures (2 past and 1 future events). Information from these sessions was used to create 1 criticism scenario related to the future and 2 related to the past, one of the latter was processed into a treatment scenario. Each of the 3 scenarios consisted of a memory anticipation part that required recalling 3 images one after another: the image of self, the surroundings, and the person of the critic involved in the scene. In the treatment scenario immediately after the imagery of the critic the rescripting part was presented, in which: 1. therapist enters the scene and prevents the criticism 2. therapist addresses a critic and points out the child's needs 3. therapist addresses the child and acknowledges its needs 4. therapist suggests to the child to perform an activity that would meet its needs.
  Interventions: Behavioral: Imagery Rescripting
- Imagery Rescripting with memory reconsolidation disruption (ImRs-DSR) (Experimental): Before treatment each participant took part in 2 imagery sessions during which a cognitive-behavioral therapist (CBT) asked him/her to recall 3 events of being criticized for failures (2 past and 1 future events). Information from these sessions was used to create 1 criticism scenario related to the future and 2 related to the past, one of the latter was processed into a treatment scenario. Each of the 3 scenarios consisted of a memory anticipation part that required recalling 3 images one after another: the image of self, the surroundings, and the person of the critic involved in the scene. In the treatment scenario 10 minutes after the imagery of the critic the rescripting part was presented, in which: 1) the therapist enters the scene and prevents the criticism 2) the therapist addresses a critic and points out the child's needs 3) the therapist addresses the child and acknowledges its needs 4) the therapist suggests to the child to perform an activity that would meet its needs.
  Interventions: Behavioral: Imagery Rescripting with Disruption of Reconsolidation
- Imagery Exposure (IE) (Experimental): Before treatment each participant took part in 2 imagery sessions during which a cognitive-behavioral therapist (CBT) asked him/her to recall 3 event of being criticized for failures. Information from these sessions was used to create 1 criticism scenario related to the future and 2 related to the past, one of the latter was processed into a treatment scenario. Each of the 3 scenarios consisted of a memory anticipation part that required recalling 3 images one after another: the image of self, the surroundings, and the person of the critic involved in the scene. In the treatment scenario the imagery of the critic was followed by the prolonged exposure to the criticism situation.
  Interventions: Behavioral: Imagery Exposure
- Compassion-Focused Therapy Imagery Rescripting (CFT_ImRs) (Experimental): Before treatment each participant took part in 2 imagery sessions during which a cognitive-behavioral therapist (CBT) asked him/her to recall 3 event of being criticized for failures. Information from these sessions was used to create 1 criticism scenario related to the future and 2 related to the past, one of the latter was processed into a treatment scenario. Each of the 3 scenarios consisted of a memory anticipation part that required recalling 3 images one after another: the image of self, the surroundings, and the person of the critic involved in the scene. In the treatment scenario immediately after the imagery of the critic the rescripting part was presented, in which: 1) therapist expressed intention to protect the child 2) desire to reduce the child's suffering 3) explained that suffering is part of the human experience 4) provided sense of community and understanding.
  Interventions: Behavioral: Compassion-Focused Therapy Imagery Rescripting

INTERVENTIONS:
Behavioral: Imagery Rescripting — Imagery Rescripting (Regular)
  Other Names: ImRs
  Arms: Imagery Rescripting (ImRs)
Behavioral: Imagery Exposure — Imagery Exposure
  Other Names: IE
  Arms: Imagery Exposure (IE)
Behavioral: Imagery Rescripting with Disruption of Reconsolidation — Imagery Rescripting with Disruption of Reconsolidation
  Other Names: ImRs-DSR
  Arms: Imagery Rescripting with memory reconsolidation disruption (ImRs-DSR)
Behavioral: Compassion-Focused Therapy Imagery Rescripting — Imagery Rescripting in Compassion-Focused Therapy
  Other Names: CFT_ImRs
  Arms: Compassion-Focused Therapy Imagery Rescripting (CFT_ImRs)

SUMMARY:
This randomized controlled trial (RCT) examines the efficacy of Imagery Exposure (IE), Imagery Rescripting (ImRs), and Compassion-Focused Therapy (CFT) in individuals with a high fear of failure. Participants (N=220) were randomly assigned to IE, ImRs, ImRs with a 10-minute break (ImRs-DSR), or CFT-based Imagery Rescripting (CFT_ImRs). Due to funding constraints, the CFT_ImRs group included a reduced sample (N=40, targeting 30 completers).

The two-week intervention consists of four structured imagery sessions. IE involves exposure to criticism-related memories without modification. In the ImRs group memory reactivation to criticism-related memories is followed by positive reappraisal. ImRs-DSR introduces a 10-minute delay before reappraisal to enhance memory updating. CFT_ImRs incorporates Compassion-Focused Therapy (CFT) principles into reappraisal, emphasizing self-compassion.

Primary outcomes include skin conductance level (SCL) and subjective emotional responses to criticism-related (and control) memories, changes in fear of failure and dysfunctional beliefs. All these variables are assessed pre-treatment, post-treatment, and at 3- and 6-month follow-ups. Results will be analyzed separately for:

IE vs. ImRs (rescripting vs. exposure and physiological predictors), ImRs vs. ImRs-DSR (memory reconsolidation effects), IE vs. CFT_ImRs (CFT vs. exposure efficacy).

DETAILED DESCRIPTION:
This study aims to investigate the efficacy and underlying psychological mechanisms of Imagery Rescripting (ImRs), Imagery Exposure (IE), and Compassion-Focused Therapy (CFT) in individuals with high fear of failure. The project is designed as a randomized controlled trial (RCT) comparing four intervention conditions: Imagery Exposure (IE), standard Imagery Rescripting (ImRs), Imagery Rescripting with a 10-minute break (ImRs-DSR), and CFT-based Imagery Rescripting (CFT_ImRs). The addition of the CFT_ImRs condition was based on the decision to explore whether compassion-focused elements provide additional benefits in reducing criticism-related subjective and autonomic responses.

The study enrolled 220 participants, randomly assigned to one of the four groups (IE, ImRs, ImRs-DSR, CFT_ImRs) in a 3:3:3:2 allocation ratio. Due to funding limitations for CFT_ImRs, recruitment for this group has been capped at 40 participants, with the goal of obtaining a final sample of 30 subjects for the study phase. The treatment phase takes two weeks starting just after pre-treatment assessments and consisting of four treatment sessions. Each of them involves exposure to autobiographical memories of childhood criticism, presented in an audio format. The IE condition involves prolonged exposure to the criticism scene without modifications. In the ImRs condition, the reactivation of memory is followed by a positive reappraisal, where an imagined caregiver acknowledges the participant's needs. In ImRs-DSR, a 10-minute break separates the memory reactivation from the positive reappraisal, aiming to enhance memory updating by increasing memory trace destabilization. In the CFT_ImRs condition, the part aiming at positive reappraisal differs from the one used in ImRs condition by incorporating some principles of Compassion-Focused Imagery Rescripting.

Primary outcome measures include physiological arousal (skin conductance level, SCL), subjective ratings, and changes in self-reported fear of failure and dysfunctional beliefs. Treatment effects will be evaluated at pre-treatment, post-treatment, and at 3- and 6-month follow-ups. The efficacy and stability of each intervention will be assessed using renewal, reacquisition, and reinstatement paradigms, as they are known from behavioral studies.

Due to the broad scope of this study, the results will be reported separately for different comparisons, as each addresses distinct research questions:

IE vs. ImRs: Examines whether rescripting differs from exposure and how the dynamics of physiological arousal influences treatment outcomes.

ImRs vs. ImRs-DSR: Investigates whether adding a mechanism for interrupting memory reconsolidation improves the efficacy of ImRs.

IE vs. CFT_ImRs: Evaluates the efficacy of Compassion-Focused Therapy in comparison to exposure-based treatment.

This study seeks to determine whether standard ImRs is better than IE and whether ImRs-DSR or CFT_ImRs provide additional benefits in reducing criticism-related subjective and autonomic responses, and whether the dynamics of physiological arousal during imagery predicts treatment responses. The findings may contribute to optimizing imagery-based therapeutic techniques for individuals with pathological fear of failure.

Due to human error in study planning, the retrospective registration for the ImRs vs. ImRs-DSR condition has already been registered in another repository under the following code: NCT06537284.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-35
* high fear of failure
* not currently undergoing psychotherapy or psychopharmacotherapy
* no severe punitive experiences in the past

Exclusion Criteria:

* current severe affective disorders
* current severe anxiety
* current severe personality disorders
* active suicidality
* psychosis
* substance abuse

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
The Performance Failure Appraisal Inventory | Screening, 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  The Performance Failure Appraisal Inventory was used to assess fear of failure. It is a 35-item questionnaire that measures the strength of subjective beliefs about the consequences of failure. The PFAI has five subscales: fear of experiencing shame and embarrassment; fear of devaluing one's self-esteem; fear of having an uncertain future; fear of important others losing interest, and fear of upsetting important others, with scores ranging 35-175.
Subjective ratings at the end of all sessions | Pre-Treatment (TP1), during 2-weeks treatment (TP2-TP5), 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  Subjective ratings at the end of all sessions - participants were asked to evaluate each fragment of the presented scenarios according to several measures: immersion, focus, emotions (happiness, sadness, guilt, fear, anger, disgust) on a 9-point Likert scale (very low-very high), and valence (very negative-very positive), scores ranging 1-9 for each factor.
SCL recordings | Pre-Treatment (TP1), during 2-weeks treatment (TP2-TP5), 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  Skin conductance level (SCL) was collected during the audio-guided scenarios' imagery at pre-treatment, treatment, post-treatment, and follow-up sessions. SCL was acquired using Biopack MP160 EDA-MRI system, with a sampling frequency of 2000Hz. The signal was resampled into 1000Hz, then smoothed with median (100 samples), and filtered with a high-passed 1Hz filter. We calculated normalized change in SCL with equation 100✕(SCLStim-SCLbaseline/SCLbaseline), where SCLStim is the mean signal value during the stimulus and SCLbaseline is an SCL reaction during the baseline preceding the first part in each scenario (Sugimine et al., 2020). Our primary outcome was SCL during the imagery of different scenarios, separated for anticipation and hotspot parts.
Saliva sampling sAA | Pre-Treatment (TP1), 2-weeks post-treatment (TP6)
  Saliva samples were collected on pre- and post-treatment with cotton rolls. Samples were collected using cotton rolls that were chewed for 1 min and were later secured in sterile V-bottom tubes and stored at 4°C temperature upon analysis. Samples were coded and sent to the Institute of Human Genetics Polish Academy of Science where the level of alpha amylase was measured.

SECONDARY OUTCOMES:
Beck Depression Inventory | Pre-Treatment (TP1), 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  Beck Depression Inventory second edition (BDI-II) is a self-report scale using 21 items regarding the presence and strength of depression symptoms, with scores ranging 0-63.
Yale-Brown Obsessive-Compulsive | Screening, 6-month Follow-up (TP8)
  Yale-Brown Obsessive-Compulsive self-report severity scale Y-BOCS-SR a 10-item, self-report questionnaire created to evaluate OCD severity, scores ranging 0-40.
The Alcohol Use Disorders Identification Test | Screening, 6-month Follow-up (TP8)
  The Alcohol Use Disorders Identification Test AUDIT is a self-reported tool containing 10 items used to assess recent alcohol consumption, alcohol dependence symptoms, and problems related to alcohol consumption, with scores ranging 0-40.
Drug Abuse Screen Test | Screening, 6-month Follow-up (TP8)
  Drug Abuse Screen Test DAST 10 is a self-reported questionnaire to detect drug use disorders, scores ranging 0-10.
Structured Clinical Interview for DSM-5 (SCID-5-PD) | Screening
  Structured Clinical Interview for DSM-5 SCID-5-PD is a semistructured clinical interview that evaluates DSM-5 personality disorders under three clusters of A, B, and C, and other specific personality disorders. Based on positive answers to questions clinician diagnose adequate personality disorders.
M.I.N.I. Mini International Neuropsychiatric Interview | Screening
  M.I.N.I. Mini International Neuropsychiatric Interview is a short structured interview for DSM IV and ICD 10 disorders, used to assess mental disorders: major depressive disorder, dysthymic disorder, suicidality, mania, panic disorder, agoraphobia, social phobia, specific phobia, obsessive-compulsive disorder, post-traumatic stress disorder, alcohol dependence/abuse, drug dependence/abuse, antisocial personality disorder. Based on positive answers to questions clinician diagnose adequate disorders.
Liebowitz Social Anxiety Scale | Pre-Treatment (TP1), 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  Liebowitz Social Anxiety Scale (LSAS) is a 24-item scale to evaluate fear and avoidance in social situations such as social interaction, public speaking, being observed by others, eating and drinking in public, with scores ranging from 0 to 144.
Pure Procrastination Scale | Pre-Treatment (TP1), 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  Pure Procrastination Scale (PPS) is composed of 12 items, which measures three components of procrastination: decisional delay, implemental delay and delays in lateness/timeliness, with scores ranging 12-60.
Frost Multidimensional Perfectionism Scale | Pre-Treatment (TP1), 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  Frost Multidimensional Perfectionism Scale was used to assess overall perfectionism and its dimensions: Personal Standards, Organization, Concern Over Mistakes, Doubts About Actions, Parental Expectations, and Parental Criticism, with scores ranging 35-175.
Social Anxiety Disorder Scale (DSM) | Screening, 6-month Follow-up (TP8)
  Self-report dimensional scale for Social Anxiety Disorder based on DSM-5 criteria. The scale consists of 10 items measuring frequency of symptoms experienced in the last 7 days. Each item is rated on a 4-point Likert scale (0 = never, 4 = all the time). Scores range 0-40, with higher scores indicating greater symptom severity.
Agoraphobia Scale (DSM) | Screening, 6-month Follow-up (TP8)
  Self-report dimensional scale for Agoraphobia based on DSM-5 criteria. The scale includes 10 items evaluating thoughts, feelings, and behaviors associated with agoraphobic avoidance in the past 7 days. Each item is scored on a 0-4 scale. Total score range: 0-40.
Panic Disorder Scale (DSM) | Screening, 6-month Follow-up (TP8)
  10-item self-rating questionnaire based on DSM-5 criteria for Panic Disorder. The scale assesses symptom frequency over the past 7 days using a 4-point Likert scale (0-4), with total scores ranging from 0 to 40.
Generalized Anxiety Disorder Scale (DSM) | Screening, 6-month Follow-up (TP8)
  A dimensional measure for Generalized Anxiety Disorder based on DSM-5, comprising 10 items. Participants indicate how frequently they experienced each symptom during the past 7 days. Scoring is on a 4-point Likert scale from 0 (never) to 4 (all the time), with total scores ranging 0-40.
Post-Traumatic Stress Symptoms Scale (DSM) | Screening, 6-month Follow-up (TP8)
  Self-report scale assessing PTSD symptoms as defined by DSM-5 criteria. The instrument includes 10 items evaluating symptom frequency over the previous 7 days on a 0-4 Likert scale. Total scores range from 0 to 40.

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław M. Michałowski, PhD, Principal Investigator — SWPS University
Locations (1):
- Poznań Laboratory of Affective Neuroscience, Institute of Psychology, SWPS University, Warsaw, Poland, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Craske MG, Kircanski K, Epstein A, Wittchen HU, Pine DS, Lewis-Fernandez R, Hinton D; DSM V Anxiety; OC Spectrum; Posttraumatic and Dissociative Disorder Work Group. Panic disorder: a review of DSM-IV panic disorder and proposals for DSM-V. Depress Anxiety. 2010 Feb;27(2):93-112. doi: 10.1002/da.20654. PMID 20099270
- [Background] Sugimine S, Saito S, Takazawa T. Normalized skin conductance level could differentiate physical pain stimuli from other sympathetic stimuli. Sci Rep. 2020 Jul 2;10(1):10950. doi: 10.1038/s41598-020-67936-0. PMID 32616939
- [Background] Wild J, Clark DM. Imagery Rescripting of Early Traumatic Memories in Social Phobia. Cogn Behav Pract. 2011 Nov;18(4):433-443. doi: 10.1016/j.cbpra.2011.03.002. PMID 22298942
- [Background] Siegesleitner M, Strohm M, Wittekind CE, Ehring T, Kunze AE. Improving imagery rescripting treatments: Comparing an active versus passive approach. J Behav Ther Exp Psychiatry. 2020 Dec;69:101578. doi: 10.1016/j.jbtep.2020.101578. Epub 2020 Jun 9. PMID 32569854
- [Background] Schiller D, Kanen JW, LeDoux JE, Monfils MH, Phelps EA. Extinction during reconsolidation of threat memory diminishes prefrontal cortex involvement. Proc Natl Acad Sci U S A. 2013 Dec 10;110(50):20040-5. doi: 10.1073/pnas.1320322110. Epub 2013 Nov 25. PMID 24277809
- [Background] Morina N, Lancee J, Arntz A. Imagery rescripting as a clinical intervention for aversive memories: A meta-analysis. J Behav Ther Exp Psychiatry. 2017 Jun;55:6-15. doi: 10.1016/j.jbtep.2016.11.003. Epub 2016 Nov 9. PMID 27855298
- [Background] Conroy, D. E., Willow, J. P., & Metzler, J. N. (2002). Multidimensional fear of failure measurement: The performance failure appraisal inventory. Journal of applied sport psychology, 14(2), 76-90.
- [Background] Arntz A, Weertman A. Treatment of childhood memories: theory and practice. Behav Res Ther. 1999 Aug;37(8):715-40. doi: 10.1016/s0005-7967(98)00173-9. PMID 10452174
- [Background] Agren T, Engman J, Frick A, Bjorkstrand J, Larsson EM, Furmark T, Fredrikson M. Disruption of reconsolidation erases a fear memory trace in the human amygdala. Science. 2012 Sep 21;337(6101):1550-2. doi: 10.1126/science.1223006. PMID 22997340
- [Derived] Baczek J, Karkosz S, Pietruch M, Szymanski R, Michalowski JM. Imagine yourself as a little girl...-efficacy and psychophysiology of imagery techniques targeting adverse autobiographical childhood experiences- multi-arm randomised controlled trial. Front Psychol. 2026 Jan 16;16:1710963. doi: 10.3389/fpsyg.2025.1710963. eCollection 2025. PMID 41625469